CLINICAL TRIAL: NCT00881452
Title: A Phase III Randomized Double Blind Placebo Controlled Trial of CM-AT in Children With Autism
Brief Title: A Trial of CM-AT in Children With Autism
Acronym: CM-AT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Curemark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00101
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Autism
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Citric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM-AT (Active Comparator): CM-AT (Luminenz-AT)- 900mg CM-AT, pancreatic enzyme concentrate (720mg)
  Interventions: Drug: CM-AT
- Placebo (Placebo Comparator): Placebo 900mg (Sucanate (98% w/w), Citric Acid (2% w/w)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM-AT — Single unit dose powder of active substance (CM-AT) administered 3 times per day for 90 days
  Other Names: 900mg CM-AT (pancreatic enzyme concentrate, 720mg
  Arms: CM-AT
Drug: Placebo — Single unit dose powder of non-active substance administered 3 times per day for 90 days
  Other Names: 900mg (Sucanate (98% w/w), Citric Acid (2% w/w)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CM-AT is safe and effective in treating the core symptoms of autism.

DETAILED DESCRIPTION:
Autism is currently a significant cause of disability in the pediatric population. Treatment is based upon the observation that many children with autism do not digest protein. CM-AT is a proprietary enzyme that is designed as a powder taken three times a day.

ELIGIBILITY:
Inclusion Criteria:

* Meets the current Diagnostic and Statistical Manual for Mental Disorders (DSM-IV-TR) diagnostic criteria for autistic disorder (AD)

Exclusion Criteria:

* Patient weighing < 11kg (24.2 lbs.)
* Demonstrated previous allergy to porcine (pork) products
* Previous history of severe head trauma or stroke, seizure within one year of entering study or uncontrolled systemic disease
* Diagnosis of: HIV, cerebral palsy, endocrine disorder, pancreatic disease
* Within 30 days of starting the study, certain supplementation, chelation or dietary restriction (a 30 day washout period would be required for inclusion)
* Use of of any stimulant medication must be discontinued 5 days prior to entering the study.
* Subject must have a stable dose of SSRI's for at least 30 days.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evidence of changes in behavior scales associated with the core symptoms of autism | Baseline, 14 days, 30 days, 60 days, 90 days

SECONDARY OUTCOMES:
Other key measures of behavior and quality of life associated with autism | Baseline, 14 days, 30 days, 60 days, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Arnold, MD MEd., Principal Investigator — Nisonger Center Ohio State University
Locations (19):
- United States (19):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - University of California, Davis, M.I.N.D. Institute, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Lake Mary Pediatrics, Orange City, Florida
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Saint Peters University Hospital, New Brunswick, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oklahoma University Child Study Center, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Houston, Houston, Texas
  - Westside Medical, Clinton, Utah

REFERENCES:
- [Background] Caronna EB, Milunsky JM, Tager-Flusberg H. Autism spectrum disorders: clinical and research frontiers. Arch Dis Child. 2008 Jun;93(6):518-23. doi: 10.1136/adc.2006.115337. Epub 2008 Feb 27. PMID 18305076
- [Background] Xue Ming, Brimacombe M, Chaaban J, Zimmerman-Bier B, Wagner GC. Autism spectrum disorders: concurrent clinical disorders. J Child Neurol. 2008 Jan;23(1):6-13. doi: 10.1177/0883073807307102. Epub 2007 Dec 3. PMID 18056691
- [Background] Simonoff E, Pickles A, Charman T, Chandler S, Loucas T, Baird G. Psychiatric disorders in children with autism spectrum disorders: prevalence, comorbidity, and associated factors in a population-derived sample. J Am Acad Child Adolesc Psychiatry. 2008 Aug;47(8):921-9. doi: 10.1097/CHI.0b013e318179964f. PMID 18645422
- [Background] Valicenti-McDermott MD, McVicar K, Cohen HJ, Wershil BK, Shinnar S. Gastrointestinal symptoms in children with an autism spectrum disorder and language regression. Pediatr Neurol. 2008 Dec;39(6):392-8. doi: 10.1016/j.pediatrneurol.2008.07.019. PMID 19027584
- [Background] Horvath K, Perman JA. Autistic disorder and gastrointestinal disease. Curr Opin Pediatr. 2002 Oct;14(5):583-7. doi: 10.1097/00008480-200210000-00004. PMID 12352252
- [Background] Parracho HM, Bingham MO, Gibson GR, McCartney AL. Differences between the gut microflora of children with autistic spectrum disorders and that of healthy children. J Med Microbiol. 2005 Oct;54(Pt 10):987-991. doi: 10.1099/jmm.0.46101-0. PMID 16157555
- [Background] Molloy CA, Manning-Courtney P. Prevalence of chronic gastrointestinal symptoms in children with autism and autistic spectrum disorders. Autism. 2003 Jun;7(2):165-71. doi: 10.1177/1362361303007002004. PMID 12846385
- [Background] Borowitz D, Goss CH, Stevens C, Hayes D, Newman L, O'Rourke A, Konstan MW, Wagener J, Moss R, Hendeles L, Orenstein D, Ahrens R, Oermann CM, Aitken ML, Mahl TC, Young KR Jr, Dunitz J, Murray FT. Safety and preliminary clinical activity of a novel pancreatic enzyme preparation in pancreatic insufficient cystic fibrosis patients. Pancreas. 2006 Apr;32(3):258-63. doi: 10.1097/01.mpa.0000202952.10612.21. PMID 16628080
- [Background] Welch MG, Welch-Horan TB, Anwar M, Anwar N, Ludwig RJ, Ruggiero DA. Brain effects of chronic IBD in areas abnormal in autism and treatment by single neuropeptides secretin and oxytocin. J Mol Neurosci. 2005;25(3):259-74. doi: 10.1385/JMN:25:3:259. PMID 15800379